CLINICAL TRIAL: NCT02039323
Title: A Feasibility Study to Assess Protection of Vaginal and Cervical Tissues From Ex-Vivo HIV-1 Challenge Following Oral Administration of Maraviroc and Tenofovir
Brief Title: A Feasibility Study to Assess Tenofovir and Maraviroc Protection Against HIV-1 in Cervical and Vaginal Explants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Angela Kashuba, PharmD, PharmD, University of North Carolina, Chapel Hill
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 13-3940
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Healthy Adult Females
Keywords: Tenofovir; Tenofovir disoproxil; Maraviroc; Pharmacologic Actions; Anti-HIV agents; Pharmacodynamics
MeSH Terms: interventions — Tenofovir; Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Participants (Experimental): Maraviroc 600 mg + Tenofovir 600 mg
  Interventions: Drug: Tenofovir; Drug: Maraviroc

INTERVENTIONS:
Drug: Tenofovir
  Other Names: Tenofovir disoproxil fumurate; Viread
Drug: Maraviroc
  Other Names: Selzentry

SUMMARY:
The purpose of this study is to determine the feasibility of a novel method to assess antiretroviral efficacy for protection against HIV-1 infection in vaginal and cervical tissue biopsies.

DETAILED DESCRIPTION:
Participants: Six premenopausal healthy volunteer women between 18-49 years of age with an intact uterus and cervix.

Procedures (methods): Subjects will be given a single dose of two oral antiretrovirals (maraviroc 600mg/tenofovir 600 mg). Subjects will be monitored and assessed for adverse events post-dose. Subjects will be sent home and asked to return in 24 hours. 24 hours post-dose, two vaginal and two cervical biopsies will be obtained. These biopsies will then be placed in an ex-vivo culture system and exposed to HIV. Viral RNA will be measured over two days to determine whether the tissues were protected from infection. A final visit for safety will be conducted 7-14 days post-enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pre-menopausal female subjects between the ages of 18-49, inclusive, with an intact uterus and cervix. (Healthy is defined as no irregular menstrual cycles or clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests)
* All subjects must have an estimated calculated creatinine clearance (eCcr) of at least 80 mL/min by the Cockcroft-Gault formula where: eCcr (female) in mL/min = [(140 - age in years) x (weight in kg) x 0.85] / (72x serum creatinine in mg/dL).
* All subjects must have a negative serum pregnancy test at screening and negative urine pregnancy tests on days of dose administration and should be using at least one of the following methods of contraception from the screening visit through 72 hours prior to first outpatient visit (at which time the women will be asked to remain abstinent until after their follow-up visit)

  * Systemic hormonal contraceptive (oral, depot, transdermal or implant)
  * Intrauterine device placed at least 1 month prior to study enrollment
  * Bilateral tubal ligation (Sterilization)
  * Vasectomized male partners
  * Condom + Spermicide
  * Unless engaged in sexual activity with female only sex partners or abstinent for at least 3 months prior with no intention of becoming sexually active during the study period. Any history of recent or present concomitant male sex partners will be addressed and ruled out in the context of screening participants for eligibility for the protocol
* Body Mass Index (BMI) of approximately 18 to 34 kg/m2; and a total body weight > 50 kg (110 lbs).
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the trial.
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.
* Subject must have documentation of a normal pap smear within 36 months of the screening visit, no procedures for abnormal cervical/vaginal pathology in the last six months, at least one prior gynecological visit as part of subject's routine medical history. If subjects have had a gynecological exam but no history of Pap smear, a Pap smear will be completed at screening and paid for by the study.
* Subject must be willing to abstain from sexual intercourse, douching, and all intravaginal objects and products for at least 72 hours prior to first study visit until study completion.
* Subject must be HIV-1 and Hepatitis B surface antigen negative as documented on screening labs.
* Subject must not be actively involved in the conception process.
* Subject must be able to swallow pills and have no allergies to any component of the study products.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including documented drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Subjects with a history of hysterectomy, or other clinically significant surgery of the female genital tract.
* Subjects who are pregnant, possibly pregnant or lactating
* Subjects with a presence of vaginal discharge or genital bleeding at screening
* History of febrile illness within five days prior to medication dosing.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.
* A positive result for HIV.
* Active Hepatitis B infection as determined by positive Hepatitis B surface antigen (HBsAg) or Hepatitis B core antibody (HBcAb) tests (in the absence of HBsAb).
* Active Hepatitis C (HCV) infection as defined by positive HCV Ab (determined by multi-antigen EIA) and detectable Hepatitis C RNA.
* A positive test for syphilis, gonorrhea, Chlamydia, or trichomonas at screening.
* Any laboratory chemistry or hematology result Grade 2 or greater according to the Division of Allergy and Infectious Disease (DAIDS) Laboratory Grading Tables
* Treatment with an investigational drug within 4 months preceding the first dose of trial medication.
* History of regular alcohol consumption exceeding 14 drinks (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of spirits) per week.
* Use of prescription or nonprescription drugs, vitamins, and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of trial medication and unable to avoid use during the inpatient pharmacokinetic visit. As an exception, systemic hormonal methods of contraception can be continued.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Allergy to lidocaine or Monsel's solution.
* Allergy to latex.
* Abnormal pap smear in the past 12 months
* Any degree of ectopy or abnormality evident during the pelvic exam at screening.
* Any condition which, in the opinion of the investigator, is likely to interfere with follow-up or ability to take the study medication appropriately.
* Unwilling or unable to comply with the following dietary and concomitant drug restrictions in regard to study drug administration as outlined in the study procedures and prohibited medications sections.
* Subjects will not be allowed to eat or drink grapefruit containing products from 7 days prior to the first dose of trial medication until after collection of biopsy sample.
* Must refrain from taking any prescription, non-prescription, herbal, vitamin or dietary supplement within at least 7 days of the study visit through completion of the study without discussing with the study staff.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Evidence of explant infection | 2 days post-biopsy
  To determine if oral administration of tenofovir plus maraviroc can protect mucosal tissues from HIV infection in an ex-vivo HIV challenge of biopsies collected post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Angela DM Kashuba, PharmD, Principal Investigator — UNC at Chapel hill
Locations (1):
- CTRC University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States